CLINICAL TRIAL: NCT05148806
Title: Mass Evaluation of Lateral Flow Immunoassays for the Detection of SARS-CoV-2 Antibody Responses in Immunosuppressed People (The MELODY Study)
Brief Title: Mass Evaluation of Lateral Flow Immunoassays for the Detection of SARS-CoV-2 (Covid-19) Antibodies
Acronym: MELODY
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: NHS Blood and Transplant (Other Government); IPSOS (Industry); University of Nottingham (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MR/W029200/1
Record Dates: First submitted 2021-12-06; First posted 2021-12-08 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Solid Organ Transplant Recipients; Autoimmune Diseases; Haematological Malignancies
Keywords: Antibody testing; SARS-COV-2; Covid-19; Immunosuppression; solid organ transplant; haematological malignancy; blood cancer; autoimmune disease
MeSH Terms: conditions — Autoimmune Diseases; COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Solid organ transplant patients: Patients who have received a solid organ transplant and who have received at least 3 doses of Covid-19 vaccine
  Interventions: Diagnostic Test: self-administered lateral flow assays
- Rare autoimmune diseases: Patients with a rare autoimmune disease who have received at least 3 doses of Covid-19 vaccine
  Interventions: Diagnostic Test: self-administered lateral flow assays
- Blood cancer: Patients with acute myeloid and lymphoid blood cancers who have received at least 3 doses of Covid-19 vaccine.
  Interventions: Diagnostic Test: self-administered lateral flow assays

INTERVENTIONS:
Diagnostic Test: self-administered lateral flow assays — The lateral flow device to be used is the Fortress COVID-19 Total Antibody Device for the detection of IgM and IgG SARS-CoV-2 against the spike protein. The device has been evaluated for use in detecting anti-S in transplant patients and found to have a sensitivity of 92% and specificity of 95%.

SUMMARY:
DESIGN Observational epidemiological study

AIMS - To determine:

1. The proportion of immunosuppressed people who have detectable SARS-CoV-2 antibodies following a primary vaccine course (3 doses), and the demographic, disease, and treatment characteristics that influence antibody status.
2. If the detection of antibodies inversely correlates with subsequent risk of severe acute respiratory syndrome coronavirus-2 infection and/or severity of disease in immunosuppressed people.

DETAILED DESCRIPTION:
The aim of this proposal is to assess at a population level; 1) the proportion of immunosuppressed people who have detectable SARS-CoV-2 antibodies following a primary vaccine course (3 doses), and the sociodemographic, disease, and treatment characteristics that influence antibody status; 2) if the detection of antibodies inversely correlates with subsequent risk of SARS-CoV2 infection and/or severity of disease in immunosuppressed individuals.

The investigators aim to target patient groups least likely to mount an immune response to vaccination; a) solid organ transplant recipients; b) patients with a rare autoimmune disease c) patients with haematological malignancies, specifically lymphoid malignancies. The investigators will use comprehensive registries to identify and recruit patients from these groups, and utilise the existing linkages these registries already have to obtain COVID-19 outcome information.

The investigators hypothesise that a sizeable proportion of immunosuppressed people will have no detectable SARS-CoV-2 antibodies following a three vaccine doses, and that this cohort is particularly susceptible to SARS-CoV-2 infection and death.

ELIGIBILITY:
Inclusion Criteria:

Adults and young people over 12 years of age, and are classified as being part of one of the following patient groups:

1. A solid organ transplant recipient (n=12,000)
2. Patients with a rare autoimmune disease (n=12,000)
3. Patients with lymphoid malignancies (n=12,000) -

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Any adult, or young person over 12 years old, with a functioning transplant who has received at least 3 vaccines, will be eligible to participate.
  2. People with rare autoimmune diseases, many of whom are on immunosuppressants, have validated disease diagnoses, and those treated with Rituximab who are most at risk of lack of seroconversion following COVID-19 vaccination.
  3. People ≥18 years of age with a haematological malignancy who have received at least 3 vaccines will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 28411 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Willicombe, MBBS, MD, Principal Investigator — Imperial College London
Locations (4):
- United Kingdom (4):
  - NHS Blood and Transplant, Bristol
  - Imperial College, London
  - Ipsos Mori, London
  - National Disease Registration Service, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Published results — https://doi.org/10.1016/S2665-9913(23)00160-1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Solid Organ Transplant Patients | Rare Autoimmune Diseases | Blood Cancer
Started | 12342 | 8117 | 7952
Completed | 9927 | 6516 | 6593
Not Completed | 2415 | 1601 | 1359

BASELINE CHARACTERISTICS:
Groups:
- Blood Cancer-Lymphoid Malignancy: Patients with acute myeloid and lymphoid blood cancers who have received at least 3 doses of Covid-19 vaccine.
  self-administered lateral flow assays: The lateral flow device to be used is the Fortress COVID-19 Total Antibody Device for the detection of IgM and IgG SARS-CoV-2 against the spike protein. The device has been evaluated for use in detecting anti-S in transplant patients and found to have a sensitivity of 92% and specificity of 95%.
- Total: Total of all reporting groups
Arm/Group | Solid Organ Transplant Patients | Rare Autoimmune Diseases | Blood Cancer-Lymphoid Malignancy | Total
Number analyzed (Participants) | 9927 | 6516 | 6593 | 23036
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Overall age is not shown because we don't have a combined dataset for the whole cohort, so this can't be reported. Those with age not reported aren't included in any of the modelling.
  years | 60 [50 to 67] | 62 [54 to 69] | 59 [49 to 67] | NA [NA to NA] — Measure Description: Overall age is not shown because we don't have a combined dataset for the whole cohort, so this can't be reported. Those with age not reported aren't included in any of the modelling.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 16 participants did not report their gender.
  Participants
    Gender: number analyzed (Participants) | 9920 | 6509 | 6591 | 23020
    Gender: Female | 4494 | 5070 | 2971 | 12535
    Gender: Male | 5426 | 1439 | 3620 | 10485
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9268 | 5992 | 6401 | 21661
  Asian | 351 | 231 | 73 | 655
  Black | 134 | 130 | 38 | 302
  Other | 133 | 142 | 64 | 339
  Not reported | 41 | 21 | 17 | 79
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9927 | 6516 | 6593 | 23036
Total number of vaccines at time of test [Count of Participants; unit: Participants] — Self-reported data on whether 3, 4 or 5+ vaccines at time of test Population: Rows added for 3, 4, 5+ vaccines at time of test
  Participants
    3 vaccines | 2700 | 2615 | 1268 | 6583
    4 vaccines | 6046 | 3531 | 4657 | 14234
    5+ vaccines | 1181 | 370 | 668 | 2219

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants With and Without Antibodies to SARS-CoV-2
Description: 1. The proportion of with and without antibodies to SARS-CoV-2 at 21 - 90 days post three vaccine doses will be presented.
Time Frame: 21 - 90 days post 3rd vaccine
Population: Patients who have received 3 vaccines
Measure: Count of Participants; unit: Participants
Arm/Group | Solid Organ Transplant Patients | Rare Autoimmune Diseases | Blood Cancer
Number analyzed (Participants) | 2700 | 2615 | 1268
Participants
  Antibody Negative | 875 | 378 | 277
  Antibody Positive | 1825 | 2237 | 991

2. Primary Outcome: The Proportion of Participants With and Without Antibodies to SARS-CoV-2
Description: 1. The proportion of participants with and without antibodies to SARS-CoV-2 at 21 - 90 days post four vaccine doses will be presented.
Time Frame: 21 - 90 days post 4th vaccine
Population: Patients who have received 4 vaccines
Measure: Count of Participants; unit: Participants
Arm/Group | Solid Organ Transplant Patients | Rare Autoimmune Diseases | Blood Cancer
Number analyzed (Participants) | 6046 | 3531 | 4657
Participants
  Antibody Negative | 1242 | 507 | 1006
  Antibody Positive | 4804 | 3024 | 3651

3. Primary Outcome: The Incidence of Participants Having at Least One RT-qPCR Proven Infection in the 6-month Follow-up Period After 3rd or 4th Vaccine
Description: The incidence of participants having at least one RT-qPCR proven infection in the 6-month follow-up will be presented for those with and without antibodies to SARS-CoV-2 after 3rd or 4th vaccine.
Time Frame: 6-month follow-up period from registration. Reporting of this is delayed following difficulties with collection of data from national bodies.
Reporting Status: Not Posted, anticipated posting 2024-12

4. Primary Outcome: The Incidence of Participants Hospitalised Due to COVID-19 and Deaths Due to COVID-19
Description: The incidence of participants hospitalised due to COVID-19 and deaths due to COVID-19 by 6 months will be presented for those with and without antibodies to SARS-CoV-2 following 3rd or 4th vaccine
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2024-12

5. Primary Outcome: Rates of Those With and Without Antibodies to SARS-CoV-2 After 3rd or 4th Vaccine
Description: Rates of those with and without antibodies to SARS-CoV-2 after 3rd or 4th vaccine will be presented for different clinical characteristics and sociodemographic factors.
Time Frame: Antibodies at 21 - 90 days after 3rd or 4th vaccine
Population: After 3rd or 4th vaccine
Measure: Number; unit: participants who received vaccines
Arm/Group | Solid Organ Transplant Patients | Rare Autoimmune Diseases | Blood Cancer
Number analyzed (Participants) | 9927 | 6516 | 6593
participants who received vaccines
  Antibody Negative after 3 vaccines: number analyzed (Participants) | 2700 | 2615 | 1268
  Antibody Negative after 3 vaccines | 875 | 378 | 277
  Antibody Positive after 3 vaccines: number analyzed (Participants) | 2700 | 2615 | 1268
  Antibody Positive after 3 vaccines | 1825 | 2237 | 991
  Antibody Negative after 4 vaccines: number analyzed (Participants) | 6046 | 3531 | 4657
  Antibody Negative after 4 vaccines | 1242 | 507 | 1006
  Antibody Positive after 4 vaccines: number analyzed (Participants) | 6046 | 3531 | 4657
  Antibody Positive after 4 vaccines | 4804 | 3024 | 3651
  Antibody Negative after 5+ vaccines: number analyzed (Participants) | 1181 | 370 | 668
  Antibody Negative after 5+ vaccines | 193 | 37 | 83
  Antibody Positive after 5+ vaccines: number analyzed (Participants) | 1181 | 370 | 668
  Antibody Positive after 5+ vaccines | 988 | 333 | 585

ADVERSE EVENTS:
Time Frame: 6 months
Description: There were no adverse events reported.
Arm/Group | Solid Organ Transplant Patients | Rare Autoimmune Diseases | Blood Cancer
All-Cause Mortality (participants affected / at risk) | 0/9927 | 0/6516 | 0/6593
Serious Adverse Events (participants affected / at risk) | 0/9927 | 0/6516 | 0/6593
Other Adverse Events (participants affected / at risk) | 0/9927 | 0/6516 | 0/6593

LIMITATIONS AND CAVEATS:
1.Participation required self-engagement 2. We used a non-quantitative test without distinguishing between absent & very low anti-SARS-CoV-2 IgG antibody concentrations nor antigen-specific T-cell responses 3.Covariates selected for the analysis were based on data captured via the research questionnaire that were clinically appropriate 4.Data processing approvals meant a single intracohort comparison analysis wasn't possible,but similar methodology & analysis was applied to the different cohorts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT05148806/Prot_SAP_000.pdf